CLINICAL TRIAL: NCT06991283
Title: The Impact of Transcutaneous Vagus Nerve Stimulation on Cardiovascular Events in Patients With Acute Myocardial Infarction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025YS-063
Record Dates: First submitted 2025-05-19; First posted 2025-05-27 (Actual); Last update posted 2025-05-27 (Actual); Status verified 2025-05

CONDITIONS: Acute Myocardial Infarction (AMI)
Keywords: acute myocardial infarcation; inflammation; vagus nerve stimulation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): Patients in this arm will receive standard care according to the guidelines after AMI. Vagus nerve stimulation is delivered through a transcutaneous electrical nerve stimulation device by attaching an ear clip to the tragus. But no stimulation will be delivered.
  Interventions: Device: Sham (no implant)
- Stimulation Group (Experimental): Patients in this arm will receive standard care according to the guidelines after AMI. Vagus nerve stimulation is delivered through a transcutaneous electrical nerve stimulation device by attaching an ear clip to the tragus. The stimulation will be performed twice daily, each session lasting for half an hour. The stimulation times are fixed between 07:00-09:00 in the morning and 19:00-21:00 in the evening, with an interval of 12 hours between the two sessions. The device is set with a pulse width of 200 microseconds and a pulse frequency of 20 hertz. The stimulation intensity is individually adjusted to above the perception threshold and below the discomfort level of 1 milliampere.
  Interventions: Device: transcutaneous vagus nerve stimulation

INTERVENTIONS:
Device: transcutaneous vagus nerve stimulation — The stimulation times are fixed between 07:00-09:00 in the morning and 19:00-21:00 in the evening, with an interval of 12 hours between the two sessions. The device is set with a pulse width of 200 microseconds and a pulse frequency of 20 hertz. The stimulation intensity is individually adjusted to above the perception threshold and below the discomfort level of 1 milliampere.
  Arms: Stimulation Group
Device: Sham (no implant) — Vagus nerve stimulation is delivered through a transcutaneous electrical nerve stimulation device by attaching an ear clip to the tragus. But no stimulation will be delivered. The sham stimulation will be performed twice daily, each session lasting for half an hour. The stimulation times are fixed between 07:00-09:00 in the morning and 19:00-21:00 in the evening, with an interval of 12 hours between the two sessions.
  Arms: Control group

SUMMARY:
The acute mortality rate of acute myocardial infarction (AMI) reduced significantly due to emergency reperfusion and subsequent treatment strategies. However, it remains a major cause of disability and death globally. Recent studies have shown that systemic inflammation is associated with infarct size and adverse clinical outcomes after myocardial infarction. Therefore, attenuating the inflammatory response may be a therapeutic target for acute coronary syndromes and improve clinical outcomes. Preclinical and clinical data indicate that vagus nerve stimulation (VNS) plays an important role in reducing the inflammatory burden and improving myocardial ischemia. However, more clinical evidence is needed to elucidate the role of VNS in patients with acute myocardial infarction and its impact on cardiovascular events. Therefore, this study aims to investigate the effect of vagal nerve modulation intervention through a prospective, randomized controlled clinical research method.

ELIGIBILITY:
**Inclusion Criteria**

1. Age between 18 and 80 years old (including 18 and 80 years old).
2. Patients with acute myocardial infarction who have undergone revascularization of the culprit vessel within 24 hours of onset.
3. Willing to participate in this study and have signed the informed consent form.

**Exclusion Criteria**

1. Hemodynamically unstable, with cardiogenic shock, requiring medication to maintain blood pressure and heart rate.
2. Baseline systolic blood pressure <90 mmHg or diastolic blood pressure <40 mmHg.
3. Average heart rate under monitoring <50 beats per minute.
4. Patients with II or III degree atrioventricular (AV) block or sick sinus syndrome who have not had a permanent pacemaker implanted.
5. Baseline (before the use of antiarrhythmic drugs) QTc interval ≥500 ms, PR interval >280 ms.
6. Patients who are participating in other clinical studies.
7. Other reasons deemed by the investigator as unsuitable for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
The occurrence of composite cardiovascular events at 3 months | 3 months after the onset of AMI
  The composite cardiovascular events including recurrent myocardial infarction，acute heart failure, ventricular arrhythmia(ventricular tachycardia,flutter and fibrillation), cardiovascular death.

SECONDARY OUTCOMES:
The occurrence of recurrent myocardial infarction, acute heart failure, ventricular arrhythmias, embolic events, and death at 3 months. | 3 month after the onset of AMI
  Separate occurrence of recurrent myocardial infarction, heart failure, ventricular arrhythmias, cardiovascular death
Changes in left ventricular ejection fraction (EF) at 3 months. | 3 month after onset of AMI
  Left ventricular ejection fraction will be calculated by cardiac echocardiography using Simpson method
Changes in BNP, IL-6, CRP and troponin-T on day 7. | Day 7 after AMI
  Changes in BNP, IL-6, CRP and troponin-T on day 7. The changes will be calculated compared with baseline(immediate result after AMI).
Changes in the 6-minute walk test at 3 month | 3 months after the onset of AMI
  6-minute walk test will performe at Day 7 and 3 month,and changes will be calculated.

IPD SHARING:
Plan to Share IPD: No